CLINICAL TRIAL: NCT05133115
Title: Resilience School-Based Intervention in Adolescents at Risk: A Clustered Randomized Control Trial.
Brief Title: Fostering Resilience in Adolescents at Risk.
Acronym: FRAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Maria Llistosella, PhD, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02-21-160-016
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Resilience, Psychological
Keywords: Adolescent; Population at Risk; Psychological Intervention; Clinical Trials, Randomized

STUDY DESIGN:
Intervention Model Description: Eligible schools will be randomly allocated either to an intervention group or control. The clusters were school classrooms (grades 6, 7). For each grade (and 7) there will be several classrooms (clusters) depending of the schools.The randomization procedure will be performed in two steps. First, the schools will be randomly allocated either to an intervention group or control by the external researcher using computer-generated random numbers; second, the external researcher will randomize the intervention group into the different school-levels.
  According to the minimum estimated sample size (70 participants/group) and knowing that there are 25 to 30 students per classroom, we will need a minimum of three clusters (classrooms) per group.
Masking Description: No-blinded participant groups and personnel (research team).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Schools with adolescents aged 12 to 15 in a context at risk. They will follow the intervention for 6 weeks (6 sessions, once a week).
  Interventions: Behavioral: Fostering Resilience in Adolescents at Risk
- Control Group (No Intervention): Schools in the control group will be all waitlisted to receive the intervention during the following academic year should it prove effectiveness. They will fill in the same research questionnaires as the Intervention group and at the same time period (January to December 2022).

INTERVENTIONS:
Behavioral: Fostering Resilience in Adolescents at Risk — The FRAK training was developed according to ecological framework, empirical evidence and contextual information. The contents, components, pedagogy, and technical elements of FRAK were established based on The Individual & Environmental Resilience Model (IERM). Previous to the intervention, a systematic review and a meta-analysis on Resilience Interventions were performed.
  Students will follow a training consisting of six 55-minute sessions: (1) introducing resilience, (2) self-esteem, (3) emotional strategies regulation, (4) social skills, (5) solving problems (6) community resources, social and peers' support.
  Other Names: FRAK
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to assess the effectiveness of a school-based resilience intervention in adolescents and to understand whether the school training can improve levels of resilience or psychological wellbeing, while reducing depressed mood.

DETAILED DESCRIPTION:
Background Some studies with adolescents reported the impact of Coronavirus disease 2019 (COVID-19) pandemic on the mental health. In the literature, resilience was related with positive mental health and was defined by some authors as a good mental health and a good psychosocial functioning despite exposure to risk or adversity (Collishaw et al., 2016). Additionally, resilience was also considered important to develop interventions to prevent or treat mental disorders, particularly anxiety, depression, and stress. Schools have been identified as one of the key settings for promoting resilience among children and young populations in this time of COVID-19 pandemic, where social inequalities have become even more evident and depressive symptoms have increased. The purpose of this trial is to assess the effectiveness of a resilience school-based intervention in adolescents and to understand whether the school training can improve levels of resilience or increase psychological wellbeing, while reducing depressed mood.

Hypothesis: Adolescents at risk between 12 and 15 years of age who receive a resilience school-based intervention by school nurses, will obtain higher scores on scales of resilience with respect to the control group, just after the intervention and 6-month post-intervention

Method:

The study is a cluster randomized controlled trial (RCT). Schools that want to participate, will sign an agreement to participate in the project Schools will be randomly allocated in control and intervention groups by external researcher using a computer-generated random numbers.

The intervention will be carried out during the school period (January to June 2022), by primary health care nurses who are part of the committee of experts and the research team. Students will follow a specific training consisting of six 55-minute sessions, once a week.

The data collection will start in January 2022 and will finish in December 2022.

Data will be collected at baseline before the intervention (T1), after 6 weeks post- intervention (T2) and 6 months after intervention as follow-up (T3).

The evaluation of the effectiveness of the intervention will be carried out using the psychometric scale CYRM-32 (as the primary outcome) which will allow us to determine changes in resilience.

Using SD of the primary outcome CYRM-32 scale, minimum sample size was calculated to be 70 students in each group, using GRANMO (https://www.imim.es/ofertadeserveis/software-public/granmo/). A follow-up loss rate of 10% was estimated.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 15 in a context of risk ( risk of social exclusion; COVID -19 pandemic context)

Exclusion Criteria:

* Adolescents aged 12 to 15 who do not want to participate in the activities of the intervention.
* Aged <12 years or >15 years

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 674 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Child Youth Resilience Measure -32 | Time 1 baseline, Time 2 post-intervention at week 6 and time 3 up to 6 months
  Changes in level of resilience using the scale Child Youth Resilience Measure -32 (CYRM-32)
  Child Youth Resilience Measure -32 (CYRM-32) The CYRM-32 includes 32 items is designed to assess resilience in children and young people (aged 12 to 23 years). It is a self-reported measure and for each question, participants use a 5-point Likert scale (1= not at all to 5= a lot (Llistosella et al., 2019).
Brief Resilience Scale | Time 1 baseline, Time 2 post-intervention at week 6 and up to 6 months
  Changes in level of resilience using the Brief Resilience scale.

SECONDARY OUTCOMES:
Emotional Regulation Strategies | Time 1 baseline, Time 2 post-intervention at week 6 and time 3 up to 6 months
  Emotion Regulation Questionnaire (ERQ) The ERQ is a self-report questionnaire, adapted in Spain by Cabello et al. (2013). It will be used to assess two emotion regulation strategies: cognitive reappraisal (6 items) and expressive suppression (4 items). Participants will answer using a 7-point Likert scale (1= strongly disagree, 7= strongly agree).
Depression Mood | Time 1 baseline, Time 2 post-intervention at week 6 and time 3 up to 6 months
  Item "Are You Depressed or Sad?" This item will assess the depression mood of the participants. It was adapted from the "Are you depressed?" Screening for depression in the terminally ill (Chochinov et al., 1997) and it is evaluate through numeric scale of 0-10 (0-not depressed, 10-worst possible depression).

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - School Antoni Ubach, Terrassa, Barcelona
  - School Goya, Terrassa, Barcelona
  - School Mediterrania, Barcelona
  - School IES Can Roca, Terrassa
  - School INS Terrassa, Terrassa
  - School Pere Viver, Terrassa
  - School Torre del Palau, Terrassa
  - School Vedruna, Terrassa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabello, R., Salguero, J. M., Fernández-Berrocal, P., & Gross, J. J. (2013). A Spanish adaptation of the Emotion Regulation Questionnaire. European Journal of Psychological Assessment, 29(4), 234-240.
- [Background] Chochinov HM, Wilson KG, Enns M, Lander S. "Are you depressed?" Screening for depression in the terminally ill. Am J Psychiatry. 1997 May;154(5):674-6. doi: 10.1176/ajp.154.5.674. PMID 9137124
- [Background] Collishaw S, Hammerton G, Mahedy L, Sellers R, Owen MJ, Craddock N, Thapar AK, Harold GT, Rice F, Thapar A. Mental health resilience in the adolescent offspring of parents with depression: a prospective longitudinal study. Lancet Psychiatry. 2016 Jan;3(1):49-57. doi: 10.1016/S2215-0366(15)00358-2. Epub 2015 Dec 2. PMID 26654748
- [Background] Limonero JT, Tomas-Sabado J, Gomez-Romero MJ, Mate-Mendez J, Sinclair VG, Wallston KA, Gomez-Benito J. Evidence for validity of the brief resilient coping scale in a young Spanish sample. Span J Psychol. 2014;17:E34. doi: 10.1017/sjp.2014.35. PMID 25012574
- [Background] Llistosella M, Gutierrez-Rosado T, Rodriguez-Rey R, Liebenberg L, Bejarano A, Gomez-Benito J, Limonero JT. Adaptation and Psychometric Properties of the Spanish Version of Child and Youth Resilience Measure (CYRM-32). Front Psychol. 2019 Jun 28;10:1410. doi: 10.3389/fpsyg.2019.01410. eCollection 2019. PMID 31316419
- [Derived] Llistosella M, Castellvi P, Garcia-Ortiz M, Lopez-Hita G, Torne C, Ortiz R, Guallart E, Una-Solbas E, Carlos Martin-Sanchez J. Effectiveness of a resilience school-based intervention in adolescents at risk: a cluster-randomized controlled trial. Front Psychol. 2024 Oct 22;15:1478424. doi: 10.3389/fpsyg.2024.1478424. eCollection 2024. PMID 39502155